CLINICAL TRIAL: NCT04707521
Title: Application of Ship - Shaped Adhesive Tape Fixing in Patients Undergoing Tracheal
Brief Title: Application of Ship - Shaped Adhesive Tape Fixing in Patients Undergoing Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2018-144
Record Dates: First submitted 2020-06-17; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: The Fixation Mainly Plays a Firm Role in the Tracheal Intubation and Reduces the Occurrence of Complications

STUDY DESIGN:
Intervention Model Description: 3M tape ship-shaped combined with strap fixing method
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3M tape ship-shaped combined with strap fixing method (Experimental): 1. Cutting method of 3M adhesive tape of ship shape: cut a piece of 20cm×3cm elastic adhesive tape, fold it in half to form a rectangle of 10cm×3cm, cut 5cm straight line from the middle point of the crease, cut it at an Angle of 45°, fold and open the 3M elastic adhesive tape in half, which is the adhesive tape required for fixing. The final shape is similar to that of a ship, and it is named as 3M adhesive tape of ship shape.
  2. Fixation method: The ship shape with 3M adhesive tape was pasted upward on the opposite cheek (near zygomatic), and the endotracheal intubation was wound around for two rounds and then glued to the near cheek (near zygomatic).Put the tooth pad next to the endotracheal intubation and wrap the tooth pad and catheter together for two turns with a short 3M adhesive tape of 12cm×1.5cm.Finally, fasten it with a lacing.
  Interventions: Behavioral: 3M tape ship-shaped combined with strap fixing method
- traditional X-shaped tape and string fixing (No Intervention): traditional X-shaped tape and string fixing

INTERVENTIONS:
Behavioral: 3M tape ship-shaped combined with strap fixing method — During fixation, the endotracheal intubation and dental pad were located in the center of the mouth, and one end of one piece of medical cloth adhesive was pasted on the patient's cheek near the side. When it reached one side of the mouth, the endotracheal intubation and dental pad were wound around twice, and then the other side of the adhesive tape was pasted on the cheek opposite the side from the other side of the mouth,The other is fixed in reverse with the same sticking method, and the two pieces of adhesive tape are finally crossed and fixed at the corners of the mouth.Finally, fasten it with a lacing
  Arms: 3M tape ship-shaped combined with strap fixing method

SUMMARY:
In order to evaluate the safety and value of the improved ship-shaped fixing on tracheal intubation patients and provide theoretical basis for clinical therapy, we conducted this research to compare the fixed effectiveness, complications, nursing workload and medical expenses about application of ship-shaped adhesive tape fixation on patient undergoing tracheal intubation.

DETAILED DESCRIPTION:
the fixed effectiveness：Incidence of catheter displacement，Incidence of unplanned extubation.

complications：Incidence f skin damage，Oral care effect，Incidence of ventilator-associated pneumonia.

nursing workload:Oral care is time-consuming medical expenses :Material economic cost

ELIGIBILITY:
Inclusion Criteria:

* Patients with SICU intubation had been intubated for <8h at the time of entry (the interval of oral care was 8h);
* Patients with brain diseases or septic shock caused by abdominal infection;
* There was no pulmonary infection before endotracheal intubation.
* Facial skin integrity;
* Good oral cavity: no odor, no residue, no oral diseases, oral mucosa integrity;
* Informed consent is given by the family members and the informed consent is signed;
* No adhesive tape allergy.

Exclusion Criteria:

* Oral injury caused by suction;
* Endotracheal intubation time < 48 h;
* In the experiment is not willing to carry on the experiment, quit voluntarily.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
the fixed effectiveness of endotracheal intubation | 34 weeks
  The tube displacement rate,

SECONDARY OUTCOMES:
Complications associated with endotracheal intubation fixation | 34 weeks
  Unplanned extubation,the occurrence of facial adhesive related skin injury,Effect of oral care

OTHER OUTCOMES:
Economic indicators | 34 weeks
  The cost of the tape required for the fixation
Nursing workload | 34 weeks
  Oral care takes a few minutes

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China